CLINICAL TRIAL: NCT04586361
Title: Prospective Analysis of Introperative RegenLab PRP and Hyaluronic Acid in Patients With Knee ACL Tear
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yi Ping Wei, Chief resident, Orthopedics department, Kaohsiung Veterans General Hospital; Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200527-2
Record Dates: First submitted 2020-09-13; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: PRP; ACL; Hyaluronic Acid
Keywords: PRP; ACL reconstruction
MeSH Terms: interventions — Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Experimental): Intraoperative1 kit of Platelet-rich plasma(PRP) injection into knee joint after anterior cruciate ligament (ACL) reconstruction.
  Interventions: Combination Product: RegenLab PRP
- Experimental group 2 (Experimental): Intraoperative1 kit of PRP+Hyaluronic acid(HA) injection into knee joint after ACL reconstruction.
  Interventions: Combination Product: hyaluronic acid
- Experimental group 3 (Placebo Comparator): Intraoperative 20 ml normal saline injection into knee joint after ACL reconstruction.
  Interventions: Other: normal saline

INTERVENTIONS:
Combination Product: RegenLab PRP — PRP preparations also improved functional outcome scores compared to hyaluronic acid and placebo in patients affected by knee osteoarthritis (OA). Based on previous studys, we can conclude that the PRP treatment is a safe and efficacious procedure which can provide functional benefit.
  Arms: Experimental group 1
Combination Product: hyaluronic acid — Few studies investigated the effects of HA+PRP combined treatment for knee osteoarthritis (OA). Numerous studies demonstrated the efficacy of HA injection therapy in knee OA for a clinical point of view, reducing the pain and improving the quality of life.
  Other Names: RegenLab PRP
  Arms: Experimental group 2
Other: normal saline — In this study, we compare introperative PRP/PRP+HA/normal saline in ACL reconstruction patient.
  Arms: Experimental group 3

SUMMARY:
Purpose: The purpose of this article is to examine the clinical application of PRP and PRP+hyaluronic acid in disorders in the knee.

Methods:

The study was conducted on 150 adult patients with age over 20 years old affected by unilateral ACL complete tear and receiving ACL reconstruction. We divided the patients in three groups, and we treated the group A with perioperative injection of HHA, group B with perioperative HHA+PRP, group C with perioperative normal saline.

Follow-up:

Every 1,3,and 12months, we recheck physical exmianation at OPD and recheck MRI at postoperative 3 months.

ELIGIBILITY:
Inclusion Criteria:

* receiving unilateral ACL reconstruction in our hospital
* postoperative follow-up over 3 month

Exclusion Criteria:

* postoperative follow-up less than 3 month
* possible pregnency
* with coagulation disease
* NSAIDs intake during study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
150 of participants with preoperative and postoperative physical examination are accessed by anterior drawer test and Lachman test | postoperative 1 month
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
150 of participants with preoperative and postoperative physical examination are accessed by anterior drawer test and Lachman test | postoperative 3 months
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
150 of participants with preoperative and postoperative physical examination are accessed by anterior drawer test and Lachman test | postoperative 12 months
  the investigators recheck physical exmianation of participants at OPD; physical examination was checked by one orthopedist
150 of participants with preoperative and postoperative Magnetic Resonance Imaging are accessed | postoperative 3 month
  anterior cruciate ligament was accessed by MRI T1 and T2 image; MRI was checked by one orthopedist

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ping Wei, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung, Taiwan